CLINICAL TRIAL: NCT04495907
Title: COVID-19 Progression in End-Stage Kidney Disease
Acronym: COPE
Status: Completed | Type: Observational
Sponsor: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-M-0047-00
Record Dates: First submitted 2020-07-30; First posted 2020-08-03 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2 Infection (Asymptomatic); SARS-CoV-2 Infection (Symptomatic)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * SARS-CoV-2 IgG
  * Genomic testing will be performed on participants with positive anti-SARS-CoV-2 IgG and/or with history of positive SARS-CoV-2 PCR results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group I- Asymptomatic patients with SARS-CoV-2 Infection
- Group II: Group II-Symptomatic patients with SARS-CoV-2 Infection

SUMMARY:
The purpose of this study is to collect genomic and clinical data among a cohort of hemodialysis patients and analyze the association between genetic markers and the development and severity of illness in response to SARS-CoV-2.

DETAILED DESCRIPTION:
COVID-19 is a novel illness caused by the SARS-CoV-2 virus. It was declared as a global pandemic on March 11, 2020 and since that time there have been outbreaks on every continent except for Antarctica. Preliminary understanding of the virus suggests that some fraction of the population does not manifest clinical disease in response to infection, others manifest a relatively benign course of illness, and still others develop a fulminant course that eventuates in the need for intensive care, mechanical ventilation, or even death. The genetic and epigenetic basis for differential susceptibility remains unknown.

Patients receiving hemodialysis provide a good opportunity to understand genetic and epigenetic susceptibility to SARS-CoV-2. By virtue of their ongoing requirements for care, such patients cannot shelter at home or maintain social distancing, but must instead report to a clinical care setting on a thrice weekly basis. Moreover, such patients often travel to and from dialysis using shared ride services, which furthers opportunity for exposure. Preliminary estimates suggest that rates of SARS-CoV-2 positivity are 2 to 5-fold higher among hemodialysis patients than in the general public. Furthermore, frequent contact with the health care system among dialysis patients makes tracking clinical course comparatively easy.

The purpose of this study is to collect genomic and clinical data among a cohort of hemodialysis patients and analyze the association between genetic markers and the development and severity of illness in response to SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older at the time of consent
* Ability to provide informed consent.
* Is currently receiving hemodialysis treatment for end-stage kidney disease at a DaVita dialysis center.
* Enrollment in prior genomics study (Additional criteria for type B only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type A & B participants must meet all of the following criteria:
  1. Is between 18 and 80 years of age, inclusive.
  2. Ability to provide informed consent.
  3. Is currently receiving hemodialysis treatment for end-stage kidney disease at a DaVita dialysis center.
  3.2 Additional Inclusion Criteria: Type B (prior participant in genomics study)
  Type B participants must meet all of the above criteria and the following criteria:
  1. Enrollment in prior genomics study.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 IgG | An average of 6 months
Anti-SARS-CoV-2 IgG | An average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Connaire, MD, Principal Investigator — Davita Clinical Research
Locations (11):
- United States (11):
  - DCR Victorville, Victorville, California
  - DCR Connecticut, Bridgeport, Connecticut
  - DCR Twin Cities, Minneapolis, Minnesota
  - DCR Las Vegas, Las Vegas, Nevada
  - DCR Bronx, The Bronx, New York
  - DCR Canton, Canton, Ohio
  - DCR El Paso, El Paso, Texas
  - DCR Lewisville, Lewisville, Texas
  - DCR San Antonio, San Antonio, Texas
  - DCR Norfolk, Norfolk, Virginia
  - DCR Milwaukee, Milwaukee, Wisconsin